CLINICAL TRIAL: NCT03140007
Title: Diagnostic Accuracy of ERCP-guided Versus Cholangioscopy-guided Tissue Acquisition in Patients With Indeterminate Biliary Strictures Suspected to be Intrinsic - a Randomized Controlled Study
Brief Title: Diagnostic Accuracy of ERCP-guided Versus Cholangioscopy-guided Tissue Acquisition in Patients With Indeterminate Biliary Strictures Suspected to be Intrinsic .
Acronym: Cholangioscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other); Evangelisches Krankenhaus Düsseldorf (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Consultant Gastroenterologist, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: AIG-002
Record Dates: First submitted 2017-04-25; First posted 2017-05-04 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Cholangiocarcinoma; Biliary Stricture
Keywords: ERCP; cholangioscopy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: prospective, multi-center, randomized controlled, post market study
Who Masked: Participant
Masking Description: prospective, multi-center, randomized controlled, post market study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm - ERCP arm (Other): Control arm- If a patient is randomized to the Control arm, then the procedure will consist of the following: ERC with recording of ERC-based impression of malignancy .ERC-guided biopsies will be collected, consisting of 6 macroscopically visible biopsies. The biopsy forceps / brush will be selected per investigator preference. ERC-guided brushing will be performed, consisting of 10 through-and-fro passes through the target lesion. After this a biliary stent will be placed under ERC-guidance if needed. A biliary sphincterotomy will be performed as needed
  Interventions: Device: ERCP guided brushing and biopsy
- Study arm - cholangioscopy arm (Active Comparator): If patient is randomized to the Study arm, then the procedure will consist of the following in order: Cannulation and sphincterotomy per standard of practice. POCS with recording of POCS-based impression of malignancy (yes/no/indeterminate). POCS will be performed using the Spy DS system. POCS-guided biopsies will be collected, consisting of 6 macroscopically visible biopsies. The POCS-guided biopsy forceps will be the SpyBite forceps.
  Interventions: Device: single operator cholangioscopy

INTERVENTIONS:
Device: single operator cholangioscopy — If patient is randomized to the Study arm, then the procedure will consist of the following in order: Cannulation and sphincterotomy per standard of practice. POCS with recording of POCS-based impression of malignancy (yes/no/indeterminate). POCS will be performed using the Spy DS system. POCS-guided biopsies will be collected, consisting of 6 macroscopically visible biopsies. The POCS-guided biopsy forceps will be the SpyBite forceps.
  Arms: Study arm - cholangioscopy arm
Device: ERCP guided brushing and biopsy — • If patients are randomized to the Control arm, then they will undergo an ERCP. ERCP-based impression of malignancy (yes/no/indeterminate) will be recorded. ERCP-guided brushing and ERCP-guided biopsy will be performed.
  Arms: Control arm - ERCP arm

SUMMARY:
Primary Objective: To assess the diagnostic accuracy of cholangioscopy-based assessment using SpyDS technology compared to cholangiography-based assessment using ERCP-guided biopsy and brushing in patients with indeterminate biliary strictures in the setting of cholangiocarcinoma.

DETAILED DESCRIPTION:
Study Design : Prospective,multi-center, randomized controlled, Post market Study (PMS)

Two groups:

* Control arm - ERCP arm: ERCP impression and ERCP-guided brushing and biopsy
* Study arm - Cholangioscopy arm: SpyDS impression and SpyDS-guided SpyBite biopsy Randomization 1:1 ratio. Primary Endpoint: Diagnostic accuracy of cholangioscopy or cholangiography assessed at 6 months after initial ERCP procedure
* Malignancy will be determined by cytology or histology on tissue sampling during the index procedure, or from other tissue acquisition or surgical specimen histopathology up to 6 months after the index procedure.
* Overall diagnostic accuracy.
* The assessed strictures will be considered benign if there was no confirmation of malignancy by 6 months after the index procedure.
* Overall diagnostic accuracy will be assessed for
* ERCP impression of malignancy
* ERCP-guided brushing and biopsies separately and combined*
* SpyDS impression of malignancy
* SpyBite biopsies
* In case of discordant results, the following will be followed for the combined pathology/cytology measure:
* If at least one is malignancy, then combine metric is malignant
* If both are benign or one is benign and one is non-diagnostic, then combined metric is benign
* If both are non-diagnostic, then combined metric is non-diagnostic

Secondary Endpoints:

1. Occurrence and severity of procedure related serious adverse events from index procedure through 30 days after procedure. Hospitalization and ICU admissions
2. Technical success of procedure defined as ability to collect tissue deemed adequate for cytology or histology. Indeterminate or equivocal or atypical or non-conclusive cytology or histology will be considered failures to this endpoint.
3. Correlation between impression of malignancy and cytopathology in the ERCP arm compared to the Cholangioscopy arm.
4. Additional diagnostic accuracy metrics: Sensitivity, specificity, positive predictive value, negative predictive value. The assessed strictures will be considered benign if there was no confirmation of malignancy by 6 months after the index procedure.
5. Impact of ERCP or cholangioscopy on patient management.
6. Need for additional diagnostic procedures beyond the index procedure.
7. Procedural measures: Type and number of devices used,
8. Duration of procedure from duodenoscope in to duodenoscope out

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older.
2. Willing and able to comply with the study procedures and provide written informed consent to participate in the study
3. Biliary obstructive symptoms
4. Indeterminate biliary stricture suspected to be intrinsic based on prior imaging

Exclusion Criteria:

1. Contraindications for endoscopic techniques
2. Prior ERCP for assessment of indeterminate biliary stricture
3. Pancreatic head mass identified on prior non-invasive imaging and thought to be the cause of the biliary obstructive symptoms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2018-02-15 (Estimated); Study Completion 2018-06-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of cholangioscopy or cholangiography | 6 Months
  Malignancy will be determined by cytology or histology on tissue sampling during the index procedure, or from other tissue acquisition or surgical specimen histopathology up to 6 months after the index procedure.The assessed strictures will be considered benign if there was no confirmation of malignancy by 6 months after the index procedure. • Overall diagnostic accuracy will be assessed for ERCP impression of malignancy, ERCP-guided brushing and biopsies separately and combined, SpyDS impression of malignancy and SpyBite biopsies

SECONDARY OUTCOMES:
Occurrence and severity of procedure related serious adverse events | 30 days
  Occurrence and severity of procedure related serious adverse events from index procedure through 30 days after procedure.
Technical success of procedure | 30 days
  Technical success of procedure defined as ability to collect tissue deemed adequate for cytology or histology. Indeterminate or equivocal or atypical or non-conclusive cytology or histology will be considered failures to this endpoint
Additional diagnostic accuracy metrics: Sensitivity, specificity, positive predictive value, negative predictive value. | 6 months
  Additional diagnostic accuracy metrics: Sensitivity, specificity, positive predictive value, negative predictive value. The assessed strictures will be considered benign if there was no confirmation of malignancy by 6 months after the index procedure
Impact of ERCP or cholangioscopy on patient management. | 6 months
  Number of patients in whom management plan is altered based on ERCP or cholangioscopy will be determined
Number of patients needed additional diagnostic procedures beyond the index procedure for final diagnosis | 6 months
  Need for additional diagnostic procedures beyond the index procedure will be noted
Number of accessories used | At index procedure.
  The total number of accessories used during the procedure in both arms will be determined.
Duration of procedure from duodenoscope in to duodenoscope out | At index procedure
  Duration of procedure is defined as time from duodenoscope in to duodenoscope out
Correlation between impression of malignancy and cytopathology in the ERCP arm compared to the cholangioscopy arm | 6 months
  Number of participants will be compared for outcome of visual impression ( benign/ malignant disease) on ERCP or cholangioscopy with final out come of cytopathology in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Ramchandani, MD DM, Principal Investigator — Asian Institute of Gastroenterology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerges C, Beyna T, Tang RSY, Bahin F, Lau JYW, van Geenen E, Neuhaus H, Nageshwar Reddy D, Ramchandani M. Digital single-operator peroral cholangioscopy-guided biopsy sampling versus ERCP-guided brushing for indeterminate biliary strictures: a prospective, randomized, multicenter trial (with video). Gastrointest Endosc. 2020 May;91(5):1105-1113. doi: 10.1016/j.gie.2019.11.025. Epub 2019 Nov 25. PMID 31778656